CLINICAL TRIAL: NCT02120625
Title: Technical Efficacy of a Direction Specific Radiofrequency Device in the Performance of Lumbar Medial Branch Neurotomies - an MRI and EMG Confirmation Study
Brief Title: Technical Efficacy of a Direction Specific Radiofrequency Device in the Performance of Lumbar Medial Branch Neurotomies
Status: Completed | Type: Observational
Sponsor: Nimbus Concepts, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: NimbusConcepts - LRFNV
Record Dates: First submitted 2014-04-20; First posted 2014-04-23 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Low Back Pain
Keywords: radiofrequency ablation; neurotomy; facet joint; medial branch; low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lumbar MB RFN: Patients undergoing lumbar medial branch radiofrequency ablation using the Nimbus MEE Probe who undergo MRI and EMG validation testing of efficacy of intended lesion production.
  Interventions: Device: Lumbar MB RFN

INTERVENTIONS:
Device: Lumbar MB RFN — Patients will be placed in a prone position and prepped. The C-arm will be adjusted to establish a true anteroposterior image of the target vertebra. The C-arm will then be rotated until the target point at the base of the SAP is clearly visualized. The Nimbus probe, with the tines (filaments) in the retracted position, will be inserted and advanced to the bony target site using a down the beam approach. The probe hub will be rotated to accomplish a full deployment of the tines with a medial or lateral angular bias, as dictated by the SAP anatomy and angle of entry of the NMEE probe. Motor stimulation at 2 Hz up to 2 volts will be administered (safety check). The lesion site will be anesthetized before the radiofrequency (RF) generator is set to achieve a temperature of 80°C for 80 seconds, following 30 second temperature ramp up. Impedance and power will be recorded.
  Other Names: Nimbus Electrosurgical Radiofrequency Multitined Expandable Electrode (MEE); Model NIM17-100-10BB

SUMMARY:
The purpose of this study is to document the effectiveness of the Nimbus Multi-tined Expandable Electrode (MEE) Probe in carrying out the heating and ablation (cutting) of the small medial branch nerves that carry pain information from the facet joints. Subjects will be selected, by way of clinical evaluation and response to medial branch blocks, to undergo this procedure of radiofrequency ablation/neurotomies of the medial branches to the specific painful facet joints of the low back in order to relieve pain. This will be carried out with an FDA-approved device using a standard technique that has been accepted throughout the world. The difference in this study is that we will make use of MRIs to image the lesion that is produced and a special EMG study to look at the muscles in the back to document the effectiveness of the device in creating the intended lesion. No other study of this kind has been produced to look at this or any other radiofrequency device in the treatment of low back pain.

DETAILED DESCRIPTION:
Study Timeline, Outline, and Methods

1. Initial evaluation with physician and study eligibility determination
2. Presentation of study to patient and informed consent obtained
3. Baseline paraspinous muscle EMG performed
4. MB (medial branch)/DR (dorsal ramus) radiofrequency neurotomy with Nimbus MEE probe (start date)
5. Post-operative soreness managed with oral and topical medications and possibly 1-4 physical therapy sessions, as needed
6. MD visit at intake evaluation and at 3 and 6 weeks following the procedure.
7. Paraspinal needle electromyography, using the mini-paraspinal mapping ("miniPM") technique of Haig will be carried out at baseline (pre-procedure) and between 3 and 6 weeks post-procedure.
8. MRI, with sequencing which allows for volumetric calculations (see Appendix III), will be obtained on all of the ten chosen subjects at 7 days post-procedure. If there is any evidence of edema or coagulation changes with volume of greater than 600 cubic mm, or evidence of bony edema or other changes believed to be due to the procedure, then a follow up MRI will be obtained at 14 days post-procedure. If bony edema changes are present at 14 days, repeat MRI will be obtained at 6 weeks post-procedure.
9. Procedural details, including procedural and fluoroscopy times, will be collected for each subject. A matched cohort of patients who have undergone MB RFN (radiofrequency neurotomy) using the previous/current method have had the same data obtained for group comparisons.

Lumbar Paraspinal Mapping:

The adequate cauterization of the targeted medial branches will be confirmed using the paraspinal mapping (PM) technique of Haig. This testing will be carried out on all subjects at 3-6 weeks post radiofrequency neurotomies, by electromyographers blinded to the side and levels of the procedure. Subjects found to have reliable evidence of spontaneous electrical activity, as detailed in, will be deemed to have had a successful denervation of the medial branch in question.

Baseline PM will also be carried out at enrollment to document a normal baseline and to rule out the presence of spontaneous activity from other underlying pathology. Those found to have findings of spontaneous activity, upon baseline needle EMG of the lumbar paraspinals, will be excluded from the study.

Lumbar MRI - Post-Procedure

The ten study participants in this study will undergo lumbar MRI, using sequencing that will allow volume calculations of any soft tissue or bony findings of edema or coagulation. Experience thus far would indicate that the zone of edema can be identified, but that the zone of tissue coagulation (smaller than the zone of edema) cannot be reliably demarcated. Bench research using the Nimbus MEE probe indicates a zone of coagulation of 550 cubic mm or less, and the expected findings on MRI would consist of a zone of edema in this range, although MRI evidence of edema may be found in a larger volume of soft tissue, given that edema changes would be expected to be present in an area larger than the area of coagulation. The intention is to provide evidence that the area treated includes the known location of the targeted medial branch, but that bone edema or other unintended findings are not encountered. These MRIs will be obtained at 7 days post-procedure. If there is evidence for unintended bony edema, then these subjects will return for repeat MRI at 14 days post-procedure. If any of these unexpected findings are still present at 14 days post-procedure, then these subjects will be asked to undergo a third MRI at 6 weeks post-procedure. Images will be interpreted by a radiologist who is board certified in diagnostic radiology. Post-procedure MRI scoring will include documentation of the presence or absence of lesions, calculated volume of lesions, whether the lesion covers the anatomical location of the medial branch, and whether there is any evidence of bone edema at the lesion site(s).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a low back pain episode greater than three months in duration, unresponsive to non-interventional care, have had a lumbar MRI which is available for review, who have been selected to undergo lumbar medial branch RF lesioning and who have agreed to undergo pre and post procedure EMG and post procedure lumbar magnetic resonance imaging (LMRI).
* Age 18 or greater
* Appropriately selected patients using at least one set of diagnostic medial branch blocks

Exclusion Criteria

* Inability to attend EMG, MRI assessments within the defined assessment time windows
* Radicular pain or evidence of neurological compromise in the lower limbs (see clarification above - Target Population).
* Those unable to read English and complete the informed consent process
* Spondylolysis or lytic spondylolisthesis, degenerative spondylolisthesis which is Grade II+ or unstable.
* Systemic inflammatory, toxic, corticosteroid induced or congenital myopathy, or inflammatory arthritis
* Possible pregnancy or other reason that precludes the use of fluoroscopy, MRI, or EMG
* Significant lumbar scoliosis (Cobb angle > 15 degrees).
* Radicular/neurological deficits or focal disc herniation and/or stenosis, with correlating radicular symptoms (defined as pain or paresthesias below the knee; pain reproduction with straight leg raising; leg > back pain with extension/rotation maneuvers; radicular strength, reflex, or sensory changes consistent with their level of nerve root impingement).
* Immunologically suppressed, or has received steroids at any dose daily for > 1 month within last 12 months
* Currently involved in another study or treatment that may affect the outcome of this study
* Evidence of spontaneous activity (denervation potentials) on baseline EMG

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Appropriate study subjects will be identified, upon initiation of care (MD/DO). They will have pain of greater than three months duration, within the current pain episode. They will have no radicular/neurological deficits or focal disc herniation and/or stenosis, with correlating radicular symptoms. They will not have any known history of ongoing radiculopathy, prior epidural spinal injections relieving their current pain, or prior lumbar surgery. These prospective patients will then undergo diagnostic medial branch blocks to determine if they are appropriate candidates for radiofrequency neurotomies and, furthermore, might also be candidates for study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Back Pain Specialists, LLC, Greenwood Village, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lumbar MB RFN
Started | 8
Completed | 6
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: adults from USA
Arm/Group | Baseline Demographics
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Magnetic Resonance Imaging (MRI) Evidence of Tissue Ablation/Edema at Targeted Lumbar Medial Branches
Description: Documentation of Magnetic Resonance Imaging (MRI) evidence of tissue ablation/edema at targeted lumbar medial branches as they course around the superior articular process and transverse process juncture of the vertebrae
Time Frame: 7 days
Population: Patients undergoing lumbar medial branch radiofrequency ablation using the Nimbus MEE Probe who undergo MRI and EMG validation testing of efficacy of intended lesion production. EMG of lumbar multifidi for medial branch lesion documentation was carried out and percent of successful lesions recorded and analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Lumbar MB RFN
Number analyzed (Participants) | 6
percentage of participants | 100

2. Primary Outcome: Volume of Lesions Were Recorded by the Reading Radiologists
Description: Volume of lesions were recorded by the reading radiologists, including proximity to medial branches
Time Frame: 7 days
Measure: Mean (95% Confidence Interval); unit: cubic millimeters
Arm/Group | Lumbar MB RFN
Number analyzed (Participants) | 6
cubic millimeters | 602 [523 to 681]

3. Primary Outcome: EMG Evidence of Lesion of the Targeted Medial Branches
Description: EMG evidence of lesion of the targeted medial branches (Percentage of positive lesions)
Time Frame: 3-6 weeks post radiofrequency ablation
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Lumbar MB RFN
Number analyzed (Participants) | 6
Number analyzed (Lesions) | 34
percentage of lesions | 88 [77 to 99]

4. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Time Frame: Up to 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lumbar MB RFN
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: 2 years, 2 months
Arm/Group | Lumbar MB RFN
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Key sub-I who performed paraspinous EMG became very ill and could not continue, and the sponsor limited funding and desire to continue after 6 reported subjects had completed their involvement in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has final say on publication of data, after their review.

Abstract of data from first 6 cases published:

Bainbridge JS, et al; Pain Medicine 2015, Volume 16, Number 8, p.1650